CLINICAL TRIAL: NCT02692612
Title: Effects of Power-velocity Muscle Characteristics During Ageing
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s58633
Record Dates: First submitted 2015-11-04; First posted 2016-02-26 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Young
- Middle-Aged
- Old

SUMMARY:
The purpose of this project is to investigate the age-related differences in force-velocity muscle characteristics during isolated knee extensions variable in speed and load, during cyclic movements on a usual and recumbent bike variable in speed and velocity development and a functional test battery with healthy participants aged between 20-80 years.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers age 20 to 80 years

Exclusion Criteria:

* Knee or hip prothesis
* Systematic training
* Cardiovascular disease
* Acute lower back pain
* Acute knee pain
* Dementia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: young (20-40y) middle-aged (40-60y) old (60-80y)
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Differences in power-velocity characteristics during ageing | 1x at baseline (cross sectional study)
  peak power and rate of power development (slope) at different velocities during knee extension movement and cyclic multijoint leg press movement compared between young and old people

SECONDARY OUTCOMES:
Reliability of strength tests on regular and recumbent bike. | 1x at baseline (cross sectional study)
  reliability of peak power and rate of power development outcomes measured twice within a period of 2 weeks
Differences in muscle fascicle characteristics during ageing. | 1x at baseline (cross sectional study)
  Differences between young and old people of fascicle shortening velocity during dynamic leg press movements measured via dynamic ultrasound
Differences in muscle activation during ageing. | 1x at baseline (cross sectional study)
  Differences in muscle activation pattern during dynamic leg press movements measured via muscle electromyography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of kinesiology and rehabilitation sciences, Leuven, Belgium